CLINICAL TRIAL: NCT02737215
Title: Prevention of Atrial Fibrillation After Coronary Artery Bypass Grafting in Patients With Obstructive Sleep Apnea: a Multicenter Study
Brief Title: Prevention of Atrial Fibrillation After Coronary Artery Bypass Grafting in Patients With Obstructive Sleep Apnea
Acronym: PAFOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rodrigo Pinto Pedrosa (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Pinto Pedrosa, MD, PhD, University of Pernambuco
Organization: University of Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAFOS01
Record Dates: First submitted 2016-04-10; First posted 2016-04-13 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP group (Active Comparator): patients will receive CPAP therapy for the first 7 days after extubation from CABG
  Interventions: Device: CPAP
- Control Group (No Intervention): Patients will receive usal care

INTERVENTIONS:
Device: CPAP — patients will receive CPAP therapy with Auto-CPAP
  Arms: CPAP group

SUMMARY:
Background. Atrial fibrillation is one of the most common complications in the postoperative period of coronary artery bypass grafting (CABG) surgery and usually associated with increased length of hospital stay and higher hospital costs. Among the main mechanisms involved, excessive sympathetic activation, oxidative stress and inflammation are fundamental elements in the pathophysiology of obstructive sleep apnea. Objectives. To evaluate the effects of continuous positive airway pressure (CPAP) in reduction of atrial fibrillation after CABG in patients with obstructive sleep apnea. Methodological procedures: A multicenter randomized controlled study to compare the incidence of atrial fibrillation between the intervention group and the control group, both monitored seven days with Holter.

ELIGIBILITY:
Inclusion Criteria:

* apnea-hypopnea index > 15 events/hour

Exclusion Criteria:

* ejection fraction < 45%
* chronic atrial fibrillation
* periprocedural instability (haemodynamic, neurological)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
atrial fibrillation | first 7 days after CABG
  will be verified by holter monitoring

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Pronto Socorro Cardiológico de Pernambuco - Procape, Recife, Pernambuco
  - Instituto de Medicina Integral Prof Fernando Figueira - Imip, Recife, Pernambuco
  - INCOR - Instituto do Coração da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chalegre ST, Barros MM, Silva BPG, Furlan SF, Giampa SQC, Marques JN, Albuquerque ALT, Monteiro VS, Drager LF, Pedrosa RP. Impact of Continuous Positive Airway Pressure on Postoperative Atrial Fibrillation in Patients with Obstructive Sleep Apnea Undergoing Coronary Artery Bypass Graft Surgery: An Exploratory Randomized Multicenter Study. Am J Respir Crit Care Med. 2022 Aug 1;206(3):358-360. doi: 10.1164/rccm.202112-2669LE. No abstract available. PMID 35549838